CLINICAL TRIAL: NCT02209155
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Phase 2 Study to Evaluate the Safety and Efficacy of R-Verapamil in the Prophylaxis of Episodic Cluster Headache
Brief Title: R-Verapamil for the Prophylaxis of Episodic Cluster Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Center Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-Verapamil-001
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Episodic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Verapamil; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-verapamil 75 mg tablet (Active Comparator): 375 mg/day; one in the morning, two in the afternoon and two at bedtime daily
  Interventions: Drug: R-verapamil 75 mg tablet
- Placebo (Placebo Comparator): one in the morning, two in the afternoon and two at bedtime daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R-verapamil 75 mg tablet
  Arms: R-verapamil 75 mg tablet
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded, randomized, parallel, placebo-controlled phase 2 study to evaluate the safety and efficacy of R-verapamil in the prophylaxis of episodic cluster headache.

DETAILED DESCRIPTION:
Approximately 30 subjects (about 15 per treatment group),will be enrolled and randomized to receive either R-verapamil or placebo for 2 weeks. The study will consist of a 1-week run-in period and a 2-week treatment period (R-verapamil or placebo). The total duration of the study for each treatment group is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman between the ages of 18 and 65
* In good health as determined by medical history and medical examination
* Has a diagnosis of episodic cluster headache as defined by the International Classification of Headache Disorders (2nd edition)
* Has a lifetime prevalence of at least 2 prior cluster bouts - Subjects must experience at least 7 attacks/week during the run-in baseline period
* Subjects must have a typical cluster period lasting at least 1 month. Subjects must be present in active cluster period and the expected remaining duration of the cluster cycle must be at least 3 weeks from Baseline Day 1 visit
* Able to differentiate other headache types from cluster headaches
* Is using or agrees to use a medically acceptable form of contraception(female of child-bearing potential)
* Negative urine pregnancy test prior to study entry(female of child-bearing potential)
* Concomitant medication that, in the opinion of the investigator and the patient's general practitioner(GP), do not pose an unacceptable risk based upon the prescribing information for verapamil
* Able to understand and comply with all study requirements
* Written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability
* Use of any drug or having any medical condition which might interact adversely with, or interfere with the action of, the study medication
* The concomitant use of beta blockers
* The consumption of grapefruit juice
* Allergic to or has shown hypersensitivity to verapamil or agents similar to verapamil
* Abuses opioids or has a history of significant drug or alcohol abuse within the past year as determined by investigator
* Has participated in an investigational drug trial in the 30 days prior to the screening visit
* Has liver or kidney disease
* Has a cardiopathology contraindicating verapamil administration
* Subjects with previous adynamic ileus.
* Subjects with chronic cluster headache
* Use of antipsychotic, antidepressants, lithium or other prophylactic treatment less than one month prior to inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in the average daily frequency of attacks | 2 weeks

SECONDARY OUTCOMES:
Change in the average daily frequency of attacks | 1 week
Change in intensity of attacks | 2 weeks
Change in duration of attacks | 2 weeks
Change in consumption of abortive agents | 2 weeks
Patient acceptability of treatment | 2 weeks
Change in headache severity index | 2 weeks
Change in Hit-6 disability score | 2 weeks
R-verapamil and Placebo responders | 2 weeks

OTHER OUTCOMES:
Adverse events assessments | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UCLH/UCL NIHR Clinical Research Facility, London, United Kingdom